CLINICAL TRIAL: NCT01115478
Title: Malaria in Pregnancy: Nutrition and Immunologic Effects
Acronym: MAL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Chair, Department of Global Health and Population, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD57941-01A2
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Malaria; Low Birth Weight; Anemia; Perinatal Mortality
Keywords: Malaria; Low birth weight; Anemia; Perinatal mortality; Vitamin A; Zinc
MeSH Terms: conditions — Malaria; Anemia; Perinatal Death | interventions — Vitamin A; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin A (Active Comparator)
  Interventions: Dietary Supplement: Vitamin A
- Zinc (Active Comparator)
  Interventions: Dietary Supplement: Zinc
- Vitamin A + Zinc (Active Comparator)
  Interventions: Dietary Supplement: Vitamin A; Dietary Supplement: Zinc
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin A — Daily oral dose of 2500 IU from enrollment until delivery
  Arms: Vitamin A; Vitamin A + Zinc
Dietary Supplement: Zinc — Daily oral dose of 25 mg from enrollment until delivery
  Arms: Vitamin A + Zinc; Zinc
Other: Placebo — Daily oral dose from enrollment until delivery
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of zinc and/or vitamin A supplementation in reducing the risk of placental malaria and its associated adverse pregnancy outcomes.

DETAILED DESCRIPTION:
Malaria accounts for a major proportion of the disease burden in Tanzania with 14 to 18 million new malaria cases being reported each year resulting in 100,000-125,000 deaths. Malaria results in impaired productivity for those between 15-55 years and lost learning opportunities in the 5-25 year age group. Dar es Salaam is characterized as an area with endemic and perennial malaria, with transmission occurring during the entire year. P. falciparum accounts for more than 95% of malaria infections. A number of interventions have contributed to reducing the burden of the disease in some settings in Tanzania and beyond, including vector control measures, bed nets, and prophylaxis and treatment of malaria. However, malaria remains a serious problem among pregnant women and children. We will examine the efficacy of micronutrient supplements as a means of enhancing immune response to malaria in pregnancy and reducing the risks of associated adverse clinical outcomes. If successful, such a low-cost intervention would be added to the armamentarium against this disease.

NOTE: The time frames listed for the maternal malaria and hemoglobin outcomes were updated on 4/22/15. This record initially indicated that maternal malaria anemia and hemoglobin would be measured at several specific time points throughout the study. Instead, maternal malaria was measured throughout pregnancy and hemoglobin was measured only at delivery. Due to an oversight, we did not update this record when this protocol change took effect at the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida or secundigravidae
* At or before 13 weeks of gestation
* HIV-negative
* Intend to stay in Dar es Salaam until delivery and for at least 6 weeks thereafter

Exclusion Criteria:

* Not primigravida or secundigravidae
* After 13 weeks of gestation
* HIV-positive
* Do not intend to stay in Dar es Salaam until delivery and for at least 6 weeks thereafter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of placental malaria | Delivery
  Placental infection status will be categorized as infected if there are asexual parasites in the placenta blood; not infected if the placental blood smear is negative; or status unknown if no placental smear is available.
Low birth weight | Delivery
  Low birth weight will be defined as birth weight less than 2500 grams.

SECONDARY OUTCOMES:
Maternal anemia | Delivery
  Anemia is defined as hemoglobin less than 11 g/dl. Severe anemia is less than 8.5 g/dl.
Perinatal death | at or after 28 weeks of gestation and in the first 7 days of life
Maternal malaria | During pregnancy
  Maternal malaria will be defined as fever within the last 72 hours with any parasitemia on a peripheral blood smear.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Ferdinand Mugusi, MD, MMed, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Muhimbili University of Health And Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Yang J, Wang D, Darling AM, Liu E, Perumal N, Fawzi WW, Wang M. Methodological approaches to imputing early-pregnancy weight based on weight measures collected during pregnancy. BMC Med Res Methodol. 2021 Feb 5;21(1):24. doi: 10.1186/s12874-021-01210-3. PMID 33546607